CLINICAL TRIAL: NCT04609124
Title: the Effect of Intravenous Metochlopramide Prophylaxis on Gastric Volume and Antral Cross Sectional Area in Patients Awaiting for Caesarean Section :a Randomized Double Blind Study.
Brief Title: Effect of Intravenous Metochlopramide Prophylaxis on Gastric Volume
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esam Hamed, Consultant, Assiut University
Other Study IDs: DASH1001
Record Dates: First submitted 2020-09-03; First posted 2020-10-30 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Aspiration Prophylaxis
Keywords: metoclopramide; cesarean section; ultrasound; gastric volume

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group:: Patients (n=35) fasting for 8 hours and received 10 mg metoclopramide intravenously diluted in 10 mL saline 0.9%.
  Interventions: Diagnostic Test: Abdominal ultrasound evaluation of antral area
- Control group:: Patients (n=35) fasting for 8 hours and received intravenous 10 mL saline 0.9% as placebo
  Interventions: Diagnostic Test: Abdominal ultrasound evaluation of antral area

INTERVENTIONS:
Diagnostic Test: Abdominal ultrasound evaluation of antral area — ultrasound assessment of antral cross sectional area
  Other Names: Nausea and vomiting episodes

SUMMARY:
Gastric fluid volume and pH in patients undergoing cesarean section are essential considerations for general anesthesia (GA). Increased gastric volume and low pH of gastric contents could predispose the risk of aspiration pneumonitis. The present study explored the research question "whether prophylaxis with intravenous metoclopramide significantly reduces gastric volume and antral cross-sectional area in patients awaiting cesarean section under GA

DETAILED DESCRIPTION:
Since regional anaesthesia has largely replaced general anaesthesia, the risk of aspiration pneumonitis during caesarean sections has significantly decreased. Nevertheless, prophylaxis against gastric aspiration is still important in patients in whom regional anaesthesia is contraindicated or in whom general anaesthesia has to be administered (for example; during emergency caesarean delivery). The administration of intravenous anaesthetics reduces the level of consciousness of a patient that compromises the protective reflexes of the upper airways. Moreover, a high level of sedation also reduces the tone of the LES (lower oesophageal sphincter). Both these situations predispose the risk of aspiration pneumonia in patients awaiting surgical interventions in supine position under general anaesthesia.

The risk of aspiration increases in outpatients if the volume of the gastric contents increases beyond 25 ml and its pH falls below 2.5. However, the risk of aspiration significantly decreases in "fasted" outpatients. Since most patients awaiting elective surgery remains fasted, routine prophylaxis for preventing aspiration pneumonitis is not recommended anymore.

the administration of intravenous metoclopramide and cimetidine across patients (n=20) awaiting laparoscopic gynaecological surgery significantly increased the pH of the gastric contents in the intervention group compared to their control counterparts (6.1 versus 2.7, p<0.05). The mean aspirated volumes were also significantly lower in the intervention group compared to their age-matched controls (6.9ml versus 15.3ml, p<0.05). Hong (2006) further showed that the percentage of individuals with high-risk gastric volume (>25 ml) and low pH (<2.5) was higher in individuals who did not receive intravenous metoclopramide and cimetidine prior to surgery compared to their counterparts who received such interventions (20% versus 5%, p<0.05) .

ELIGIBILITY:
Inclusion Criteria:

* pregnant women belonging to the age range between 22 to 38 years and who provided informed consent to participate.

Exclusion Criteria:

* a neurological and psychological disorders
* renal or hepatic diseases
* chronic gastroesophageal reflux diseases
* refusal to consent

Ages: 22 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Study Population: pregnant females
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2021-10-24 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
effect of S intravenous metoclopramide prophylaxis on gastric volume | 2 hours
  antral cross section will be measured using ultrasound machine before and after metoclopramide injection

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
only the outcome of the study no personal identity will be revealed